CLINICAL TRIAL: NCT05429229
Title: Effect of Combined Antioxidant Therapy in Eye Drops on Inflammatory and Oxidative Stress Biomarkers in Tear Film in Patients With Diabetic Retinopathy and Dry Eye Syndrome
Brief Title: Effect of Topical Antioxidants in Dry Eye Disease and Diabetic Retinopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adolfo Daniel Rodriguez-Carrizalez (Other)
Collaborators: Hospital Civil de Guadalajara (Other)
Responsible Party: Sponsor-Investigator, Adolfo Daniel Rodriguez-Carrizalez, Principal Investigator, University of Guadalajara
Organization: University of Guadalajara (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSRD-20200831-1
Record Dates: First submitted 2022-05-30; First posted 2022-06-23 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Dry Eye Syndromes; Diabetic Retinopathy; Oxidative Stress; Tear Film Deficiency
Keywords: Dry Eye Disease; Oxidative Stress biomarkers; Inflammatory biomarkers; Tear film; Eye drops; Diabetic Retinopathy
MeSH Terms: conditions — Dry Eye Syndromes; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Clinical trial phase 2 A.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Q10 coenzyme, vitamin E and cross-linked hyaluronic acid (Experimental): This arm will administer eye drops with a combination of cross-linked hyaluronic acid, Q10 coenzyme and vitamin E, it will consist of 26 patients with diabetic retinopathy and mild to moderate dry eye syndrome. One drop will be instilled in each eye every 4 hours for a month.
  Interventions: Drug: VisuXL®
- Sodium hyaluronate (Active Comparator): This arm will administer eye drops with sodium hyaluronate, it will consist of 26 patients with diabetic retinopathy and mild to moderate dry eye syndrome. One drop will be instilled in each eye every 4 hours for a month.
  Interventions: Drug: Lagricel PF®
- Sodium hyaluronate and chondroitin sulfate (Active Comparator): This arm will administer eye drops with a combination of sodium hyaluronate and chondroitin sulfate, it will consist of 26 patients with diabetic retinopathy and mild to moderate dry eye syndrome. One drop will be instilled in each eye every 4 hours for a month.
  Interventions: Drug: Humylub PF®

INTERVENTIONS:
Drug: VisuXL® — It consists of a preservative-free eye drop composed of 100 mg cross-linked hyaluronic acid, 100 mg coenzyme Q10, 500 mg vitamin E TPGS (D-alpha-tocopheryl polyethylene glycol succinate), one drop is applied in each eye every 4 hours for a month.
  Other Names: VisuXL tear drop
  Arms: Q10 coenzyme, vitamin E and cross-linked hyaluronic acid
Drug: Lagricel PF® — It consists of a preservative-free eye drop composed of sodium hyaluronate 0.4%, one drop is applied in each eye every 4 hours for a month.
  Other Names: Lagricel preservative free
  Arms: Sodium hyaluronate
Drug: Humylub PF® — It consists of eye drops without preservatives composed of 0.1% sodium hyaluronate and 0.18% chondroitin sulfate, one drop is applied to each eye every 4 hours for a month.
  Other Names: Humylub preservative free
  Arms: Sodium hyaluronate and chondroitin sulfate

SUMMARY:
The main objective of our study is to evaluate the effect of eye drops with antioxidants on mild to moderate dry eye symptoms in patients with diabetic retinopathy, evaluating the levels of inflammatory cytokines and oxidative stress in the tear film.

The researchers intend to include 78 patients, divided into three intervention groups, who will be randomly assigned an eye drop with antioxidants, where the patient must apply one drop in each eye for 1 month.

In the study, the characteristics of the surface of the eye will be evaluated and tear samples will be taken from each eye, before and after the intervention with the eye drops. Subsequently, the clinical and sample results will be evaluated to compare the effects between them.

DETAILED DESCRIPTION:
Dry eye syndrome is a multifactorial disease where tear film homeostasis is lost, accompanied by ocular symptoms such as burning, blurred vision, foreign body sensation, ocular redness, itching, in which tear film instability and hyperosmolarity, causing inflammation of the ocular surface, endothelial damage and neurosensory alterations.

Worldwide, in patients with diabetic retinopathy it has a prevalence of 54%, however in Mexico, only a prevalence of 41% has been described in the diabetic population, without having reports of prevalence in patients with diabetic retinopathy.

The state of chronic hyperglycemia in diabetes mellitus causes neuropathic corneal damage and dysfunction of the meibomian glands, this promotes a decrease in tear production, establishing dysfunction of the tear film and a state of hyperosmolarity in it, the latter induces activation of inflammatory mediators and release of proinflammatory cytokines that generate more damage to the corneal surface, entering a vicious cycle of tear film instability.

Likewise, the preexisting state of oxidative stress in patients with diabetic retinopathy, where there is an imbalance between the production and degradation of reactive oxygen species, contributes to the induction of changes in the corneal surface and tear film dysfunction.

Dry eye treatment is focused on the characteristics of the tear film and the characteristics of the ocular surface, with the aim of controlling and improving symptoms, with the use of different formulations and tolerability profiles. However, these are not adequate to reduce the effect of the inflammatory state and oxidative stress present in the tear film and the ocular surface, causing the patient's visual quality to worsen.

The researchers intend to assess whether antioxidant therapy in eye drops influences levels of oxidative stress and inflammatory markers in the tear film.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes, with presence of diabetic retinopathy in any of its stages without data on severity
* Patients who voluntarily give their informed consent.
* Patients who meet an Ocular Surface Disease Index (OSDI) score between 13-32 points (mild to moderate severity)
* Patients who meet one or more of the following:
* Tear film breakup time equal to or less than 10 seconds
* Corneal fluorescein staining with more than 5 sites
* Conjunctival staining with more than 9 sites.
* Non-smokers or history of inactive smoking > 6 months
* Metabolic criteria:
* Glycated hemoglobin equal to or less than 9%
* LDL less than or equal to 100 mg/dl
* Triglycerides less than or equal to 180 mg/dl
* Blood pressure less than or equal to 140/80 mm Hg

Exclusion Criteria:

* Patients with autoimmune diseases and/or Sjögren's disease
* Patients with neurodegenerative processes and/or cancer
* Present aggregate ophthalmological diagnosis of:
* Glaucoma
* Allergic, viral or bacterial conjunctivitis.
* Demodex
* Eye parasitic infections.
* Unresolved eye trauma
* Scarring diseases of the ocular surface
* Corneal or conjunctival ulcers.
* Filamentous keratitis, neurotrophic
* Bullous keratopathy
* Patients taking any of the following medications:
* Osmotic diuretics
* Alpha agonists
* NSAIDs, cannabinoids or opioids
* Benzodiazepines, selective serotonin reputate inhibitors, monoamine oxidate inhibitors
* nonlepromatous, antimalarials (Chloroquine / Hydroxychloroquine)
* Corticosteroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in levels of tumor necrosis factor alpha (TNF-a) in tear film at 30 days. | 30 days
  Tears will be collected with Drummond glass® micro capillary tubes without stimulation of tear secretion and placed in an eppendorf tube at -80 celsius degrees. The cytokine concentration will be determined with multiplex bead immunoassays technique and reported in picogram per milliliter units (pg/mL)
Change from baseline in levels of interleukin 8 (IL-8) | 30 days
  Tears will be collected with Drummond glass® micro capillary tubes without stimulation of tear secretion and placed in an eppendorf tube at -80 celsius degrees. The cytokine concentration will be determined with multiplex bead immunoassays technique and reported in picogram per milliliter units (pg/mL)
Change from baseline in levels of interleukin 6 (IL-6) | 30 days
  Tears will be collected with Drummond glass® micro capillary tubes without stimulation of tear secretion and placed in an eppendorf tube at -80 celsius degrees. The cytokine concentration will be determined with multiplex bead immunoassays technique and reported in pg/mL.
Change from baseline in levels of interleukin 10 (IL-10) | 30 days
  Tears will be collected with Drummond glass® micro capillary tubes without stimulation of tear secretion and placed in an eppendorf tube at -80 celsius degrees. The cytokine concentration will be determined with multiplex bead immunoassays technique and reported in picogram per milliliter units (pg/mL)
Changes from baseline in total antioxidant capacity in the tear film at 30 days. | 30 days
  Tears will be collected with Drummond glass® micro capillary tubes without stimulation of tear secretion and placed in an eppendorf tube at -80 celsius degrees. Total antioxidant capacity concentration will be determined with colorimetric assay technique and reported in units called Trolox equivalents (TE), nmol/sample.
Change from baseline in lipoperoxides levels in tear film at 30 days. | 30 days
  Tears will be collected with Drummond glass® micro capillary tubes without stimulation of tear secretion and placed in an eppendorf tube at -80 celsius degrees. Lipoperoxides concentration will be determined with colorimetric assay technique and reported in nmol/mL.

SECONDARY OUTCOMES:
Change from baseline in the pattern of ocular surface staining with fluorescein sodium according to Oxford Scheme at 30 days. | 30 days
  Ocular surface staining with fluorescein sodium dye it will be assessed during slit lamp examination and it will be measure on a scale from 0 to 5 according to the Oxford scheme, with 5 being the most severe staining.
Change from baseline in the pattern of ocular surface staining with lissamine green according to Oxford Scheme at 30 days. | 30 days
  Ocular surface staining with lissamine green dye it will be assessed during slit lamp examination and it will be measure on a scale from 0 to 5 according to the Oxford scheme, with 5 being the most severe staining.
Change from baseline in the tear break-up time (TBUT) in seconds at 30 days. | 30 days
  It will be measured the time interval in seconds between a complete blink and the first appearance of a dry spot in the tear film after fluorescein sodium administration during slit-lamp examination, considering less than 10 seconds as abnormal.
Change from baseline in tear film osmolarity at 30 days. | 30 days
  It will be measured collecting a tear sample in each eye with TearLab® Test reporting osmolarity in milliosmol per liter (mOsm/L)
Change from baseline in tear secretion in mm with Schirmer I test at 30 days. | 30 days
  Tear secretion will be assessed with a graduated test strip placed on the lower eyelid margin without anesthesia, after five minutes, the strip is removed and the amount of wetting is measured in mm, less than 10 mm is considered abnormal.

OTHER OUTCOMES:
Change from baseline severity of dry eye symptoms according the punctuation in Ocular Surface Disease Index (OSDI) at 30 days | 30 days.
  OSDI is a questionnaire that will be assessed on a scale of 0 to 100 to measure dry eye disease severity (normal, mild to moderate and severe) and effect on vission-related function.

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo D Rodriguez-Carrizalez, M.D/PhD, Study Director — University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics,, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Lopez-Contreras AK, Martinez-Ruiz MG, Olvera-Montano C, Robles-Rivera RR, Arevalo-Simental DE, Castellanos-Gonzalez JA, Hernandez-Chavez A, Huerta-Olvera SG, Cardona-Munoz EG, Rodriguez-Carrizalez AD. Importance of the Use of Oxidative Stress Biomarkers and Inflammatory Profile in Aqueous and Vitreous Humor in Diabetic Retinopathy. Antioxidants (Basel). 2020 Sep 20;9(9):891. doi: 10.3390/antiox9090891. PMID 32962301
- [Background] Pastor-Maldonado CJ, Suarez-Rivero JM, Povea-Cabello S, Alvarez-Cordoba M, Villalon-Garcia I, Munuera-Cabeza M, Suarez-Carrillo A, Talaveron-Rey M, Sanchez-Alcazar JA. Coenzyme Q10: Novel Formulations and Medical Trends. Int J Mol Sci. 2020 Nov 10;21(22):8432. doi: 10.3390/ijms21228432. PMID 33182646
- [Background] Postorino EI, Rania L, Aragona E, Mannucci C, Alibrandi A, Calapai G, Puzzolo D, Aragona P. Efficacy of eyedrops containing cross-linked hyaluronic acid and coenzyme Q10 in treating patients with mild to moderate dry eye. Eur J Ophthalmol. 2018 Jan;28(1):25-31. doi: 10.5301/ejo.5001011. Epub 2018 Feb 19. PMID 28777385
- [Background] Najafi L, Malek M, Valojerdi AE, Aghili R, Khamseh ME, Fallah AE, Tokhmehchi MR, Behrouz MJ. Dry eye and its correlation to diabetes microvascular complications in people with type 2 diabetes mellitus. J Diabetes Complications. 2013 Sep-Oct;27(5):459-62. doi: 10.1016/j.jdiacomp.2013.04.006. Epub 2013 May 30. PMID 23726741
- [Background] Graue-Hernandez EO, Serna-Ojeda JC, Estrada-Reyes C, Navas A, Arrieta-Camacho J, Jimenez-Corona A. Dry eye symptoms and associated risk factors among adults aged 50 or more years in Central Mexico. Salud Publica Mex. 2018 Sep-Oct;60(5):520-527. doi: 10.21149/9024. PMID 30550113
- [Background] Gao Y, Zhang Y, Ru YS, Wang XW, Yang JZ, Li CH, Wang HX, Li XR, Li B. Ocular surface changes in type II diabetic patients with proliferative diabetic retinopathy. Int J Ophthalmol. 2015 Apr 18;8(2):358-64. doi: 10.3980/j.issn.2222-3959.2015.02.26. eCollection 2015. PMID 25938056
- [Background] Fong PY, Shih KC, Lam PY, Chan TCY, Jhanji V, Tong L. Role of tear film biomarkers in the diagnosis and management of dry eye disease. Taiwan J Ophthalmol. 2019 Sep 12;9(3):150-159. doi: 10.4103/tjo.tjo_56_19. eCollection 2019 Jul-Sep. PMID 31572651
- [Background] Seen S, Tong L. Dry eye disease and oxidative stress. Acta Ophthalmol. 2018 Jun;96(4):e412-e420. doi: 10.1111/aos.13526. Epub 2017 Aug 21. PMID 28834388
- [Background] Dogru M, Kojima T, Simsek C, Tsubota K. Potential Role of Oxidative Stress in Ocular Surface Inflammation and Dry Eye Disease. Invest Ophthalmol Vis Sci. 2018 Nov 1;59(14):DES163-DES168. doi: 10.1167/iovs.17-23402. PMID 30481822
- [Background] Navel V, Sapin V, Henrioux F, Blanchon L, Labbe A, Chiambaretta F, Baudouin C, Dutheil F. Oxidative and antioxidative stress markers in dry eye disease: A systematic review and meta-analysis. Acta Ophthalmol. 2022 Feb;100(1):45-57. doi: 10.1111/aos.14892. Epub 2021 May 2. PMID 33938134
- [Background] Rodriguez-Carrizalez AD, Castellanos-Gonzalez JA, Martinez-Romero EC, Miller-Arrevillaga G, Pacheco-Moises FP, Roman-Pintos LM, Miranda-Diaz AG. The effect of ubiquinone and combined antioxidant therapy on oxidative stress markers in non-proliferative diabetic retinopathy: A phase IIa, randomized, double-blind, and placebo-controlled study. Redox Rep. 2016 Jul;21(4):155-63. doi: 10.1179/1351000215Y.0000000040. Epub 2015 Aug 31. PMID 26321469
- [Result] Rodriguez-Carrizalez AD, Castellanos-Gonzalez JA, Martinez-Romero EC, Miller-Arrevillaga G, Villa-Hernandez D, Hernandez-Godinez PP, Ortiz GG, Pacheco-Moises FP, Cardona-Munoz EG, Miranda-Diaz AG. Oxidants, antioxidants and mitochondrial function in non-proliferative diabetic retinopathy. J Diabetes. 2014 Mar;6(2):167-75. doi: 10.1111/1753-0407.12076. Epub 2013 Aug 21. PMID 23875878